CLINICAL TRIAL: NCT04124081
Title: Pharmacokinetic Interactions Between Hydronidone and Entecavir Capsules in Healthy Chinese Subjects(Single Center, Single Arm, Open, Self - Control)
Brief Title: Pharmacokinetic Interactions Between Hydronidone and Entecavir Capsules in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GNI-F351-201503
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-04

CONDITIONS: Hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug group (Experimental)
  Interventions: Drug: Hydronidone capsules& Entecavir capsules

INTERVENTIONS:
Drug: Hydronidone capsules& Entecavir capsules — take the Hydronidone capsule and then the entecavir capsule, and then take the last two together

SUMMARY:
This study, by comparing the Hydronidone capsules and entecavir capsule in a single dose and steady-state dosing state of both the level of blood drug concentration, assess Hydronidone capsules and entecavir capsule for interaction。

ELIGIBILITY:
Inclusion criteria：

1. gender: Chinese healthy male subject;
2. age: 18-40 years old, with a difference of no more than 10 years;
3. weight: ≥50kg; Body mass index [= weight kg/ (height m2)] ranged from 19 to 24.
4. the subject (or his/her partner) has no pregnancy plan during and within 6 months after the trial and voluntarily takes effective physical contraception and has no sperm donation plan;
5. before the trial, I have had a detailed understanding of the nature, significance, possible benefits, possible inconveniences and potential risks of the trial, and I have volunteered to participate in the clinical trial. I am able to communicate well with the investigator, comply with the requirements of the whole study, and have signed a written informed consent.

Exclusion criteria：

1. have participated in any other clinical trials within the first three months of the trial;
2. (preliminary) of any process may affect test security, or drug in the body of the disease, including but not limited to: heart, liver, kidney, endocrine, the digestive tract, immune system and respiratory system always or the existing system diseases (especially cardiovascular diseases including cardiovascular disease risk, any impact on drug absorption of gastrointestinal diseases (such as irritable bowel syndrome symptoms, bowel disease or inflammatory bowel disease), active pathological bleeding (such as peptic ulcer), urticaria, eczema, dermatitis, epilepsy, allergic rhinitis, asthma, etc.);
3. (consultation) allergy: if there are two or more drugs, food allergy history (including experimental drugs), lactose intolerance;
4. (consultation) any drugs that inhibit or induce drug metabolism in the liver (common liver enzyme inducers: barbiturates (phenobarbital is the most common), carbamazepine, aminoximate, griseofulvin, aminopropyl, phenytoin, gromitol, rifampin, dexamethasone; Common liver enzyme inhibitors: ampromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide); Or have used any medicines (including Chinese herbal medicines) or health supplements within 14 days prior to initial administration;
5. (consultation) have special requirements on food and cannot follow a uniform diet (such as intolerance to standard meals) or have difficulty swallowing;
6. (consultation) unable to tolerate venipuncture and/or having a history of blood or acupuncture;
7. (consultation) patients who have been drinking excessive amounts of tea, coffee or caffeinated drinks (more than 8 cups a day, 1 cup =250mL) for a long time; Or taking any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) within 48 hours before the first administration of the drug;
8. (consultation) previous binge drinking (i.e., male drinking more than 28 units per week and female drinking more than 21 units per week (1 unit contains 14g alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or who had regularly consumed alcohol (more than 14 units per week) during the 6 months prior to the trial; Or who had taken any alcoholic product within 24 hours of initial administration;
9. (consultation) those who had donated blood or suffered massive bleeding (greater than 450 mL) within 3 months before the first administration of the study, or who planned to donate blood or blood components during the study period or within 3 months after the end of the study;
10. (consultation) acute disease during the screening phase before study or before study medication;
11. (consultation) patients who had taken food or drinks containing enzymes that can induce or inhibit liver metabolism (e.g., grapefruit, mango, pitaya, grape juice, orange juice, etc., rich in flavonoids or citrus glycosides) within 24 hours before the first administration were studied;
12. (consultation) those who have had surgery within three months before the screening period, or who are planning to have surgery during the study period, and those who have had surgery that will affect drug absorption, distribution, metabolism and excretion;
13. (consultation) previous history of drug abuse; A history of drug abuse;
14. (consultation) those who have smoked more than 5 cigarettes per day in the 14 days before screening, or who cannot stop using any tobacco products during the trial;
15. screening for smoking or using any tobacco products up to admission;
16. screening phase physical examination, measurement of vital signs, electrocardiogram examination, laboratory examination [blood routine, urine routine, blood biochemistry, blood coagulation function], and the investigator judged abnormal patients with clinical significance;
17. those with positive nicotine test results;
18. alcohol breath test with test results greater than 0.0mg/100ml;
19. positive urine drug screening;
20. hepatitis b surface antigen positive, or hepatitis c antibody positive, or syphilis spirochete antibody positive, or HIV antibody positive;
21. the investigator considers that there are any circumstances that may affect the subject's informed consent or adherence to the study protocol, or participation in the study may affect the study results or their own safety.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentration | up to 12 weeks
  Compare the difference in plasma drug concentration between single drug and two drug combinations

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics committee of drug clinical trials of huazhong university of science and technology, Wuhan, Hubei, China